CLINICAL TRIAL: NCT04686292
Title: Diagnostic Accuracy of Urine Flow Cytometry in Diagnosing and Excluding Bacteruria in the Emergency Department
Brief Title: Diagnostic Accuracy of Urine Flow Cytometry in Excluding Bacteruria
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: SHS-ED-12b-2020
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Acute Infection
Keywords: Emergency department; Acute infections; bacteruria; urinary tract infections; diagnosis
MeSH Terms: conditions — Emergencies; Urinary Tract Infections; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected infection: All patients admitted to the emergency department with suspected infections assessed by the receiving physician
  Interventions: Diagnostic Test: urine flow cytometry

INTERVENTIONS:
Diagnostic Test: urine flow cytometry — Diagnostic test of urine flow cytometry. A urine sample will be collected according to routine procedure by a study assistant. The sample will be divided into two aliquots; half for routine urine culturing, and half for Point-of-care Urine Flow cytometry (POC-UFC) analysis (UF-5000, Sysmex, Kobe, Japan). The analysis will be performed according to manufacturer's instruction and conducted by laboratory staff. Laboratory staff will be blinded to the participants diagnosis and outcome. The results of the POC-UFC analysis will not be visible to the treating physician.

SUMMARY:
A more rapid test for bacteriuria is desired. This will exclude the patients not having bacteriuria, which will contribute to a more rapid and accurate diagnosis of infectious diseases. The aim of the study is to investigate the diagnostic accuracy of point-of-care urine flow cytometry on diagnosing and excluding bacteriuria

DETAILED DESCRIPTION:
A prerequisite for the appropriate use of antibiotics is timely access to accurate diagnostic tests, since treatment of acute infections should be initiated within a few hours to avoid serious complications such as bacteremia, sepsis, organ failure, septic shock and death.

The diagnosis of urinary tract infections including acute pyelonephritis (APN) is difficult due to often weak and non-specific symptoms and high incidence of asymptomatic bacteruria in especially elderly patients. The diagnosis is verified by significant bacteriuria in urine culture.

Unfortunately, the time from urine sample to result from urine cultures is more than 24 hours days. Urine test strips are unreliable with low specificity and low predictive values. Therefore, a point-of-care (POC) test is desired, which can provide rapid results and quickly identify a bacteriuria. One such tool may be urine flow cytometry (UFC), which has shown promising diagnostic value for the exclusion of bacteriuria with a high negative predictive value. However, better documentation for its use as an ED diagnostic screening method is needed.

The aim of the study is to investigate the diagnostic accuracy of POC-UFC on diagnosing and excluding bacteriuria? Our hypothesis is that by excluding patients not having bacteriuria, it will contribute to a more rapid and accurate diagnosis

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of acute infections assessed by the receiving physician at the emergency department

Exclusion Criteria:

* If the attending physician considers that participation will delay a life-saving treatment or patient needs direct transfer to the intensive care unit.
* Admission within the last 14 days
* Verified COVID-19 disease within 14 days before admission
* Pregnant women
* Severe immunodeficiencies: Primary immunodeficiencies and secondary immunodeficiencies (HIV positive CD4 <200, Patients receiving immunosuppressive treatment (ATC L04A), Corticosteroid treatment (>20 mg/day prednisone or equivalent for >14 days within the last 30 days), Chemotherapy within 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acutely admitted patients with suspected infections from three emergency departments (EDs) in the Region of Southern Denmark (Hospital Sønderjylland, Hospital Lillebælt, Odense University Hospital)
Sampling Method: Probability Sample
Enrollment: 966 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Bacteriuria | urine collected within 4 hours of arrival to emergency department and analysed within one week
  The urine culture analysis combined with microbiologist assessment will be used as reference standard for bacteriuria. Diagnostic accuracy will be conducted, and Youden index analysis will be used to estimate the best cut-off

SECONDARY OUTCOMES:
Verified infectious diagnosis by expert panel | 2 months after discharge
  An expert panel will define the final diagnosis (including APN) based on all findings during admission. The expert panel consists of two independent consultants from the emergency department with significant experience in emergency medicine and acute infections. They will individually determine the type of infection the patient admitted actually had. The final diagnosis will be based on all available relevant information from the patient medical record including MRI of kidneys and HR-CT of lungs. A standardized template will be used. Disagreement will be discussed until a consensus is reached.

OTHER OUTCOMES:
Intensive care unit treatment | within 60 days from admission to emergency department
  transfer to ICU during current admission (binary outcome)
Length of stay | within 60 days from admission to emergency department
  days spent in hospital during current admission
The number of participants who died within 30 days | within 30 days from arrival day
  binary - 30-days mortality
The number of participants who died within 90 days | within 90 days from arrival day
  binary - 90 days mortality
Readmission | within 30 days from day of discharge
  binary
In-hospital mortality | within 60 days from admission to emergency department
  binary
Level of infection markers | blood collected within 4 hours of arrival to emergency department
  Concentration of serum procalcitonin, CRP and suPAR
Urological intervention | Measured 7 days after admission
  Number of patients, who during the course of admission with suspected acute pyelonephritis requires urological interventions

CONTACTS AND LOCATIONS:
Overall Officials: Christian Backer Mogensen, Study Chair — Hospital of Southern Jutland
Locations (1):
- Hospital of Southern Jutland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koves B, Cai T, Veeratterapillay R, Pickard R, Seisen T, Lam TB, Yuan CY, Bruyere F, Wagenlehner F, Bartoletti R, Geerlings SE, Pilatz A, Pradere B, Hofmann F, Bonkat G, Wullt B. Benefits and Harms of Treatment of Asymptomatic Bacteriuria: A Systematic Review and Meta-analysis by the European Association of Urology Urological Infection Guidelines Panel. Eur Urol. 2017 Dec;72(6):865-868. doi: 10.1016/j.eururo.2017.07.014. Epub 2017 Jul 25. PMID 28754533
- [Background] Herraez O, Asencio MA, Carranza R, Jarabo MM, Huertas M, Redondo O, Arias-Arias A, Jimenez-Alvarez S, Solis S, Zamarron P, Illescas MS, Galan MA. Sysmex UF-1000i flow cytometer to screen urinary tract infections: the URISCAM multicentre study. Lett Appl Microbiol. 2018 Mar;66(3):175-181. doi: 10.1111/lam.12832. Epub 2018 Jan 28. PMID 29223137
- [Derived] Skjot-Arkil H, Heltborg A, Lorentzen MH, Cartuliares MB, Hertz MA, Graumann O, Rosenvinge FS, Petersen ERB, Ostergaard C, Laursen CB, Skovsted TA, Posth S, Chen M, Mogensen CB. Improved diagnostics of infectious diseases in emergency departments: a protocol of a multifaceted multicentre diagnostic study. BMJ Open. 2021 Sep 30;11(9):e049606. doi: 10.1136/bmjopen-2021-049606. PMID 34593497